CLINICAL TRIAL: NCT02664896
Title: Determination of Pain Phenotypes in Older Adults With Knee Osteoarthritis
Brief Title: Pain Phenotypes in Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 12-1188
Record Dates: First submitted 2015-12-18; First posted 2016-01-27 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Osteoarthritis, Knee; Pain
Keywords: Knee pain; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — 1mL of whole blood will be taken for analysis of inflammatory factors including IL-1beta, IL-6, IL-8, TNF, and C-Reactive Protein. Samples will be stored at University of Colorado Hospital until analysis is complete. Samples will then be destroyed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Knee Osteoarthritis Cohort: Subjects with knee osteoarthritis will be asked to participate in the knee osteoarthritis testing session. This group will participate in 1 three hour testing session.
  Interventions: Other: Knee Osteoarthritis
- Healthy Subject Cohort: Healthy subjects will be asked to participate in the healthy control testing session. This group will participate in 1 two hour testing session.
  Interventions: Other: Healthy Control

INTERVENTIONS:
Other: Knee Osteoarthritis — Questionnaire completion, strength testing, gait testing, pressure-pain threshold testing, proprioception testing, knee measurements, blood draw, and knee radiographs.
  Groups: Knee Osteoarthritis Cohort
Other: Healthy Control — Questionnaire completion, strength testing, gait testing, pressure-pain threshold testing, proprioception testing, and knee measurements.
  Groups: Healthy Subject Cohort

SUMMARY:
Recently, the medical community has learned damage to the knee joint may be one of many possible reasons for pain in knee osteoarthritis. Psychological factors and other aspects of brain function seem to play an important role in the pain experience. Although research studies have examined these factors on an individual basis, no study has examined all of these factors in the same population. Furthermore, some measures of brain function- having to do with perception of the painful body part- have yet to be examined in knee osteoarthritis. The investigators plan to study many of these variables in a group of people with knee osteoarthritis, as well in some healthy controls (without knee pain), in order to establish the relative importance of these measures in contributing to pain, as well as validate new measures of perception in people with knee osteoarthritis. We also plan to use a statistical tool- known as latent profile analysis- to look at subgroups of knee osteoarthritis pain. The hypothesis is that different people experience pain in knee osteoarthritis for different reasons. This study will be the first study to use all of these different variables- which can be reproduced in a clinical setting- to look for different subgroups of knee osteoarthritis pain. Ultimately, the goal is to help clinicians better prioritize and target interventions to individual patients. The investigators believe this will lead to better outcomes and fewer treatment complications currently associates with pharmaceutical and surgical interventions that are widely used to treat knee osteoarthritis.

DETAILED DESCRIPTION:
In a 2011 statement to the Food and Drug Administration, the Osteoarthritis Research Society International (OARSI) identified the "phenotyping" of OA pain as a research priority to "better target pain therapies to individual patients." Successful identification of pain phenotypes will allow new interventions to be tested in homogeneous populations of patients presenting with similar pain pathophysiology, ultimately enhancing treatment effects in defined populations for whom interventions are determined safe and effective. Clinical populations of knee OA are clearly heterogeneous, spanning wide age ranges and encompassing patients with a wide variety of functional abilities. The pain experience in knee OA may be similarly individualized and complex; some patients may present with pain that appears attributable to classic signs of joint damage, while others may present with pain due to psychological distress or central mechanisms. Changes in somatosensory processing and pain threshold are also known to occur with aging. However, the scientific community has yet to examine these variables concurrently in the same study population. Therefore, the relative importance of each of these measures in determining pain severity across the lifespan is unknown. It is also unknown whether these variables (or interactions between variables) are representative of different pain phenotypes in knee OA. This is an important yet unresolved question; a patient with high levels of psychological distress and low levels of joint damage may warrant a different intervention strategy than the traditional knee-directed approach. On the other hand, someone with increased psychological distress in addition to severe joint damage may benefit from traditional interventions that are further augmented with other impairment-specific interventions. This sort of targeted approach is the topic of current research in other chronic pain populations, where a similar conceptual model, composed of peripheral, psychological and central components to the pain experience (among others), is recognized.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-85
* Diagnosed with Knee Osteoarthritis by a physician or by ACR clinical criteria

Exclusion Criteria:

* sensory dysfunction due to injury (i.e. known nerve damage)
* neurological diagnosis affecting sensory or motor function (e.g. stroke, Parkinson's Disease, multiple sclerosisetc.)

Healthy Volunteers eligibility criteria:

* Age 50-85
* Do not possess knee osteoarthritis diagnosis
* do not have knee pain
* do not have a history major knee trauma or lower extremity trauma or surgery
* do not have any other pain condition

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subject population will include 50-85 year olds who experience knee pain and have been diagnosed with knee osteoarthritis by a physician. Additionally, a healthy control cohort will be recruited. This cohort will also be 50-85 years old but will deny having any pain and will not be diagnosed with knee osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2013-04; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Knee Pain Measured by Visual Analog Scale (VAS) | Baseline

SECONDARY OUTCOMES:
Quadriceps Strength Testing with CSMI Humac Norm Isokinetic Dynamonmeter | Baseline
Hamstrings Strength Testing with CSMI Humac Norm Isokinetic Dynamonmeter | Baseline
Knee Range of Motion | Baseline
Girth for Swelling Measurement of Knee | Baseline
Tactile Threshold Test | Baseline
Two Point Discrimination Test | Baseline
Gait Speed Test | Baseline
Five Time Sit-To-Stand | Baseline
Pressure/Pain Threshold Test | Baseline
Pressure/Pain Threshold Test Conditioned Pain Modulation | Baseline
Laterality Recognition Test | Baseline
Perception of Limb Size Test | Baseline
Comorbidity Index | Baseline
Intermittent and Constant Osteoarthritis Pain: Knee Version | Baseline
KOOS Knee Survey | Baseline
Arthritis Efficacy Scale | Baseline
Tampa Scale for Kinesiophobia | Baseline
Pain Catastrophizing Scale | Baseline
Center for Epidemiologic Studies Depression Scale | Baseline
Inflammatory Cytokines | Baseline
  IL-1beta, IL-6, IL-8, TNF, C-Reactive Protein
Kellgren-Lawrence Grade of Knee Radiographs | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Stevens-Lapsley, PT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Background] Kittelson AJ, Stevens-Lapsley JE, Schmiege SJ. Determination of Pain Phenotypes in Knee Osteoarthritis: A Latent Class Analysis Using Data From the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2016 May;68(5):612-20. doi: 10.1002/acr.22734. PMID 26414884
- [Background] Kittelson AJ, George SZ, Maluf KS, Stevens-Lapsley JE. Future directions in painful knee osteoarthritis: harnessing complexity in a heterogeneous population. Phys Ther. 2014 Mar;94(3):422-32. doi: 10.2522/ptj.20130256. Epub 2013 Oct 31. PMID 24179141
- [Background] Brandt KD, Dieppe P, Radin EL. Etiopathogenesis of osteoarthritis. Rheum Dis Clin North Am. 2008 Aug;34(3):531-59. doi: 10.1016/j.rdc.2008.05.011. PMID 18687271
- [Background] Maillefert JF, Roy C, Cadet C, Nizard R, Berdah L, Ravaud P. Factors influencing surgeons' decisions in the indication for total joint replacement in hip osteoarthritis in real life. Arthritis Rheum. 2008 Feb 15;59(2):255-62. doi: 10.1002/art.23331. PMID 18240195
- [Background] McAlindon TE, Cooper C, Kirwan JR, Dieppe PA. Knee pain and disability in the community. Br J Rheumatol. 1992 Mar;31(3):189-92. doi: 10.1093/rheumatology/31.3.189. PMID 1540789